CLINICAL TRIAL: NCT01003548
Title: Comparison of the in Vitro Development of Human Embryos in Static and and Microfluidics Systems of Culture
Brief Title: Embryo Development in Microfluidics System of Culture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Incept Biosystems (Unknown)
Responsible Party: José Roberto Alegretti, Universidade Federal de São Paulo
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 0405/08
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Infertility
Keywords: Embryo culture; IVF; Microfluidics; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Static culture (Active Comparator): Embryos individually cultured in microdrops of 40 microliters of G-IVFplus series V
  Interventions: Device: Static culture
- Smart plataform (Experimental): Embryos culture in dynamics microfluidic culture system
  Interventions: Device: SMART dynamic system of embryo culture

INTERVENTIONS:
Device: SMART dynamic system of embryo culture — Embryos will be cultured in a dynamic system of microfluidics.
  Arms: Smart plataform
Device: Static culture — Embryos cultured in 40 microliters microdrops of G-IVF plus series V
  Arms: Static culture

SUMMARY:
Embryo culture is a cornerstone of in vitro fertilization treatments. Usually, embryos are cultured in microdrops of culture media in incubators with controlled temperature, humidity and atmosphere. However, these culture systems are static, while in vivo the initial growth of the embryo takes place in the uterine tube and they are submitted to a dynamic environment. The aim of this study is to compare the embryo development on days 2 and 3 of culture morphological features of embryos under static and dynamic(microfluidics) systems of culture.

DETAILED DESCRIPTION:
Embryo culture is a cornerstone of in vitro fertilization treatments. Usually, embryos are cultured in microdrops of culture media in incubators with controlled temperature, humidity and atmosphere. However, these culture systems are static, while in vivo the initial growth of the embryo takes place in the uterine tube and they are submitted to a dynamic environment. The aim of this study is to compare the embryo development on days 2 and 3 of culture morphological features of embryos under static and dynamic(microfluidics) systems of culture.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 35 years old
* No more than 1 previous IVF failure
* Absence of physical conditions that can interfere in oocyte quality
* At least 8 zigotes 24 hours after fertilization

Exclusion Criteria:

* Use of epididimary or testicular sperm
* Sperm or egg donation
* Untreated systemic diseases

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Embryo morphology on days 2 and 3 of embryo culture according to the criteria described by Lucinda Veeck | Embryo culture for 3 days before transference to the uterus

SECONDARY OUTCOMES:
Implantation rate and pregnancy rate | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo LA Motta, MD, PhD, Study Chair — Department of Gynecology - Universidade Federal de Sao Paulo
Locations (1):
- Departamento de Ginecologia, São Paulo, São Paulo, Brazil